CLINICAL TRIAL: NCT05319132
Title: A Phase 0 Study to Evaluate DF-003 in ex Vivo Assays Using Peripheral Blood Mononuclear Cells (PBMC) From Subjects With Retinal Dystrophy, Optic Nerve Edema, Splenomegaly, Anhidrosis and Headache (ROSAH) Syndrome.
Brief Title: Evaluate DF-003 in ex Vivo Assays Using Peripheral Blood Mononuclear Cell From Subjects With ROSAH Syndrome
Acronym: ROSAH
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0299
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Unrecognized Condition
Keywords: ROSAH Syndrome.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 blood samples of 7 ml for ex-vivo analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adult subjects with ROSAH syndrome — The main objective is to evaluate the ex vivo inhibitory potential of DF-003 on alpha-1 kinase activity.

SUMMARY:
Alpha-1 kinase (ALPK1) has been reported as a potential causative gene for ROSAH Syndrome.

Genetic variants including T237M have been found in ROSAH Syndrome patients. Our in-house study has found that T237M mutation leads to hyperactivity of ALPK1, which may be the cause of the inflammatory syndromes found in ROSAH Syndrome patients. We hypothesize that T237M mutation ALPK1 cause ROSAH Syndrome and an ALPK1 inhibitor can be a potential therapy for treating this disease. To test our hypothesis, we designed an experiment in which ex vivo peripheral blood mononuclear cells (PBMCs) from ROSAH Syndrome patients will be exposed to a potent ALPK1 inhibitor (DF-003) or placebo. We expect to see downregulation of activated inflammatory genes, chemokine/cytokines and acute phase proteins in the ROSAH Syndrome patient samples that are exposed DF-003.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 18
* Patient with ROSAH syndrome with the confirm T237M mutation

Exclusion Criteria:

* person under legal protection or under protectives measures
* person unable to express consent
* person in emergency situation (vital or not)
* person infected by Human Immunodeficiency Virus and/or Hepatitis B Virus and/or Hepatitis C Virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns adult subjects with ROSAH syndrome
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2028-05-06 (Estimated); Study Completion 2028-05-06 (Estimated)

PRIMARY OUTCOMES:
Cytokine release assays | At day 0
  The Cytokine release assays will analyzed by ELISA in cells supernatants the Interleukin 8 (IL-8), Tumor Necrosis Factor (TNF) concentrations in the presence/absence of DF-003 and control.

CONTACTS AND LOCATIONS:
Overall Officials: YVAN JAMILLOUX, Principal Investigator — Service de medecine interne - Hôpital de la Croix Rousse
Locations (5):
- France (5):
  - Hôpital Nord Croix Rousse, Lyon, Auvergne-Rhône-Alpes
  - service de Genetique - Institut de Biologie Santé PBH-IBS, Angers
  - Hôpital de la Pitié Salpétrière, Paris
  - Service D'ophtalmologie, Reims
  - Service de médecine interne et immunologie clinique, Rennes